CLINICAL TRIAL: NCT00707044
Title: Short-Stay Intensive Care for Coronary Artery Bypass Patients,Development of a Guideline for Giving Adequate Care on the Cardiosurgical Intensive Care
Brief Title: Short-Stay Intensive Care for Coronary Artery Bypass Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Health Care Insurance Board (nr: 00106), Amstelveen, The Netherlands (Unknown)
Responsible Party: Mr. M. van Essen, Dutch Health Care Insurance Board
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 01-039; 00106 (CVZ)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2008-06

CONDITIONS: Coronary Artery Bypass
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Short-Stay Intensive Care treatment (SSIC), 8 hours of Intensive care treatment
  Interventions: Procedure: Short-Stay Intensive Care treatment (SSIC)
- B (Active Comparator): control group, care as usual, 24 hours intensive care stay
  Interventions: Procedure: Control group (usual care)

INTERVENTIONS:
Procedure: Control group (usual care) — control group, care as usual, 24 hours intensive care stay
  Arms: B
Procedure: Short-Stay Intensive Care treatment (SSIC) — Short-Stay Intensive Care treatment (SSIC), 8 hours of Intensive care treatment
  Arms: A

SUMMARY:
Objective: To evaluate the safety and cost-effectiveness of Short Stay Intensive Care (SSIC) treatment for low-risk coronary artery bypass patients Design: Randomized clinical equivalence trial Setting: University Hospital Maastricht, the Netherlands Patients: low-risk coronary artery bypass patients Interventions: 600 patients were randomly assigned to undergo either SSIC treatment (8 hours Intensive Care) or control treatment (care as usual, overnight Intensive Care).

Measurements: The primary outcome measures were Intensive Care (IC) readmissions and total hospital stay. The secondary outcome measures were total hospital costs, Quality of Life (QoL), postoperative morbidity and mortality. Hospital costs consisted of the cost of hospital admission(s) and outpatient costs.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass patients

Exclusion Criteria:

* age older than 78 years,
* ejection fraction of less than 30%
* stage 3 obesity (BMI>40kg/m2)
* haemodialysis (kidney replacing therapy)
* pulmonary hypertension (systolic <40mmHg)
* recent CVA (<1month)
* recent myocardial infarction (<24hours)
* cardiogenic shock, (systolic blood pressure<80mmHg,
* central filling pressure>20mmHg,
* cardiac index<1.8 litres/minute/m2),
* need for inotropic therapy (>5mg/mcg/min. dopamine or dobutamine)
* ongoing infarction (a significant increase of enzyme "CKMB" within 4 hours before surgery)
* the need for intra-aortic balloon pump
* inability to give informed consent
* inability to speak/ read/ understand the Dutch language
* patients who had emergency surgery.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2001-01; Primary Completion 2003-10 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Intensive Care (IC) readmissions | one month postoperative

SECONDARY OUTCOMES:
total hospital stay, total hospital costs, postoperative morbidity and mortality | one month
generic and disease specific Quality of Life (QoL) | one year postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ghislaine van Mastrigt, Msc, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Result] van Mastrigt GA, Heijmans J, Severens JL, Fransen EJ, Roekaerts P, Voss G, Maessen JG. Short-stay intensive care after coronary artery bypass surgery: randomized clinical trial on safety and cost-effectiveness. Crit Care Med. 2006 Jan;34(1):65-75. doi: 10.1097/01.ccm.0000191266.72652.fa. PMID 16374158